CLINICAL TRIAL: NCT01813136
Title: A Randomized, Multicenter, Open-label, Phase II Study of the Optimal Scheme of Administration of Pazopanib in Thyroid Carcinoma
Brief Title: Phase II Study of the Optimal Scheme of Administration of Pazopanib in Thyroid Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAZOTHYR; 2012-003162-41 (EudraCT Number)
Record Dates: First submitted 2013-03-11; First posted 2013-03-18 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Thyroid Carcinoma
Keywords: radioiodine refractory Differentiated Thyroid Carcinoma; pazopanib; intermittent administration; time to treatment failure; TUTHYREF
MeSH Terms: conditions — Thyroid Neoplasms | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous pazopanib (Arm A) (Active Comparator): Daily oral administration of pazopanib 800mg (28 days cycles) from randomization until progression (according to RECIST 1.1) under treatment, after an initial period of 6 cycles (28 days) of daily administration of pazopanib 800mg from inclusion until randomization
  Interventions: Drug: Continuous pazopanib (Arm A)
- Intermittent pazopanib (Arm B) (Experimental): Temporary discontinuation of pazopanib at randomization, after an initial period of 6 cycles (28 days) of daily administration of pazopanib 800mg from inclusion until randomization. Pazopanib will be reintroduced for 6 cycles of 28 days, with daily administration of pazopanib 800mg, as soon as the patient relapses (progressive disease according to RECIST 1.1). At the end of this additional 6 cycles, study drug will be stopped a second time.
  This sequential scheme will be maintained until the patient experiences "on-treatment" progression
  Interventions: Drug: Intermittent pazopanib (Arm B)

INTERVENTIONS:
Drug: Continuous pazopanib (Arm A) — Daily oral administration of pazopanib 800mg (28 days cycles) from randomization until progression (according to RECIST 1.1) under treatment, after an initial period of 6 cycles (28 days) of daily administration of pazopanib 800mg from inclusion until randomization
  Other Names: GW786034
  Arms: Continuous pazopanib (Arm A)
Drug: Intermittent pazopanib (Arm B) — Temporary discontinuation of pazopanib at randomization, after an initial period of 6 cycles (28 days) of daily administration of pazopanib 800mg from inclusion until randomization. Pazopanib will be reintroduced for 6 cycles of 28 days, with daily administration of pazopanib 800mg, as soon as the patient relapses (progressive disease according to RECIST 1.1). At the end of this additional 6 cycles, study drug will be stopped a second time.
  This sequential scheme will be maintained until the patient experiences "on-treatment" progression
  Other Names: GW786034
  Arms: Intermittent pazopanib (Arm B)

SUMMARY:
The objective of this study is to determine the feasibility of pazopanib treatment interruption with reintroduction at progression in iodine refractory progressive Differentiated Thyroid Cancer (DTC) patients as compared to pazopanib continuous administration.

DETAILED DESCRIPTION:
Total or near-total thyroidectomy is the primary treatment for differentiated thyroid carcinoma. Postoperatively, DTC are treated with radioiodine (131I) and thyroid stimulating hormone (TSH) suppressive levothyroxine therapy.

But 5% to 20% of patients with DTC develop distant metastases; some of them become refractory to 131I therapy.

Targeted therapies have been studied in iodine refractory DTC for several years but none of these treatments has yet been approved in DTC and clinicians continue to enroll patients in clinical trials. The agents used so far in thyroid cancer are small molecules sharing the property to inhibit various tyrosine kinase receptors such as Vascular Endothelial Growth Factor Receptor (VEGFR), Epidermal Growth Factor Receptor (EGFR), RET or c-met.

The VEGF (Vascular Endothelial Growth Factor) is one of the several pro angiogenic molecules that play a pivotal role in angiogenesis, one of the mechanisms involved in tumor growth and dissemination.

VEGF expression is highly prevalent in Papillary Thyroid Carcinoma (PTCs) (79%), Follicular Thyroid Carcinoma (FTCs) (50%) or Poorly Differentiated Thyroid Carcinoma (PDTCs) (37%) and VEGFR is respectively expressed in 76%, 83% and 25% for VEGRF-1 and 68%, 56% and 37% for VEGRF-2.

Pazopanib (GW786034 - GlaxoSmithKline) is an orally administered, potent multitarget tyrosine kinase inhibitor of VEGFR in particular (but also of PDGFR-α and -β, and stem cell factor receptor c-Kit).

The results obtained in metastatic or locally advanced refractory DTC are currently available (phase II study of 39 patients with metastatic, rapidly progressive RAI-refractory DTC, treated with pazopanib 800mg daily, were published in Lancet Oncology in 2010 by KC Bible), demonstrating the efficacy of these therapies in this indication. However, no clear data is yet available indicating the optimal duration of treatment in first line therapy: patients are currently treated until progression or until drug discontinuation due to toxicity. Indeed, patients may have some difficulties to manage the chronic mild to moderate (grade 1-2) side-effects related to long-term treatment, leading some asymptomatic patients in whom tumor is controlled by TKI treatment to ask for treatment interruption.

The intermittent administration should avoid the occurrence of long-term adverse event and subsequent dose reductions or discontinuation, thus allowing a longer control of underlying disease.

All these considerations led our reflexion in the design of the present study, that is to say to determine the feasibility of pazopanib treatment interruption with reintroduction at progression in iodine refractory progressive DTC patients as compared to pazopanib continuous administration, after 6 initial cycles of pazopanib 800 mg daily for all patients included in the study, with a strong rationale for intermittent administration of pazopanib.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old,
* Histologically confirmed diagnosis of differentiated thyroid cancer (papillary, follicular and poorly differentiated)
* Archival tumor sample available. It will be provided for all subjects, for biomarker analysis before and/or during study treatment.
* Patients must have been treated with therapeutic RAI. Patients may have received prior treatment with either 1 line of chemotherapy and/or up to 1 Tyrosine Kinase Inhibitor,
* Resistance to therapeutic radioiodine (RAI) (for DTC) as demonstrated at least by one of the following:

  * Absence of iodine uptake in at least one target lesion on a post-therapy radioactive iodine scan,
  * Presence of a target lesion after a cumulative radio-iodine activity of at least 600 mCi,
  * Patient with uptake who have RAI treatment of at least 100 mCi within the last 12 months and have disease progression,
* Documented progression as per RECIST 1.1 based on 2 consecutives imaging performed within the last 12 months,
* Measurable disease according to RECIST version 1.1,
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1,
* Adequate organ system function defined as the following:

Hematology:

* Absolute Neutrophils Count (ANC) ≥ 1.5 Gi/L
* Hemoglobin ≥ 9 g/dL (5.6µM) (transfusion is not allowed within 7 days of screening assessments)
* Platelets ≥ 100 Gi/L
* Prothrombin Time (PT) ≤ 1.2 x ULN or International Normalized Ratio (INR) ≤ 1.2 Subjects receiving anticoagulant therapy are eligible if their INR is stable and within the recommended range for the desired target of anticoagulation
* Activated Partial Thromboplastin Time (aPTT) ≤ 1.2 x ULN

Electrolytes :

- Potassium within normal ranges.

Hepatic :

* Total bilirubin ≤ 1.5 x ULN
* Alanine AminoTansferase (ALAT) and Aspartate AminoTransferase (ASAT) ≤ 2.5 x ULN Concomitant elevation in bilirubin and ASAT/ALAT above 1.0xULN is not allowed

Renal :

* Serum creatinine ≤ 1.5 mg/dL (133µM) or if serum creatinine> 1.5 mg/dL, calculated creatinine clearance (ClCR) ≥ 50 mL/min (Cockcroft formula or MDRD formula for patients older than 65 years old)
* Urine Protein to Creatinine Ratio (UPC) < 1; If UPC ratio ≥ 1, then a 24-hour urine protein must be assessed. Subjects must have a 24-hour urine protein value < 1 gram to be eligible Use of urine dipstick for renal function assessment is not acceptable

  * Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days of first dose of pazopanib. They must be willing to use effective contraception methods during the study and up to 7 days after the last pazopanib administration.
  * Affiliated to the French social security system.
  * Subjects must provide written informed consent prior to perform any study-specific procedure or assessment and must be willing to comply with treatment and follow up.

Note: Procedures conducted as part of the subject's routine clinical management (e.g., blood count, imaging study such as bone scan) and obtained prior to signing of informed consent may be utilized for screening or baseline purposes provided these procedures are conducted as specified in the protocol,

Exclusion Criteria:

* Other histological sub-types of thyroid tumors like medullar carcinoma, anaplastic carcinoma, lymphoma or sarcoma,
* Prior treatment with pazopanib,
* Prior malignancy, Subjects who have had another malignancy and have been disease-free for 5 years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible
* Symptomatic metastases of Central nervous system (CNS) requiring or having required steroids or enzyme-inducing anticonvulsants within 4 weeks before inclusion ,
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

  * Active peptic ulcer disease,
  * Known intraluminal metastatic lesion with risk of bleeding,
  * Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation,
  * History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to begin study treatment,
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

  * Malabsorption syndrome,
  * Major resection of the stomach or small bowel,
* Corrected QT interval (QTc) > 480 msec (correction method according to the Bazett's method),
* History of any one or more of the following cardiovascular conditions within the past 6 months :

  * Cardiac angioplasty or stenting,
  * Myocardial infarction,
  * Unstable angina,
  * Coronary artery bypass graft surgery,
  * Symptomatic peripheral vascular disease,
  * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA),
  * Cerebrovascular accident including Transient Ischemic Attack (TIA), pulmonary embolism or untreated Deep Venous Thrombosis (DVT), Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible,
* Poorly controlled hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg) as described in the section 7.2 "Study requirements" of this protocol, Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. At least one day after antihypertensive medication initiation or adjustment, blood pressure (BP) must be re-assessed three times at approximately 2-minute intervals. These three values should be averaged to obtain the mean diastolic blood pressure and the mean systolic blood pressure. The mean SBP / DBP ratio must be <140/90 mmHg (OR 150/90 mm Hg, if this criterion is approved by the coordination center) in order to be eligible.
* Major surgery or trauma within 28 days prior to first dose of investigational product and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement are not considered to be major surgery),
* Evidence of active bleeding or bleeding diathesis,
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage, Lesions infiltrating major pulmonary vessels (contiguous tumor and vessels) are excluded; however, the presence of a tumor that is touching, but not infiltrating (abutting) the vessels is acceptable (CT with contrast is strongly recommended to evaluate such lesions).

  * Large protruding endobronchial lesions in the main or lobar bronchi are excluded; however, endobronchial lesions in the segmented bronchi are allowed.
  * Lesions extensively infiltrating the main or lobar bronchi are excluded; however, minor infiltrations in the wall of the bronchi are allowed.
* Hemoptysis within the last 8 weeks before inclusion,
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drug,
* Treatment with any of the following anti-cancer therapies :

  * radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib (analgesic radiation therapy is allowed if the radiation field doesn't include a potential target lesion for tumor assessments),
  * chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib,
* Administration of other oncologic drug or any non-oncologic investigational drug within 30 days (or 5 half lives whichever is longer) prior to receiving the first dose of study treatment, or planned to be administered during the study participation,
* Unable or unwilling to discontinue use of prohibited medications listed in Section 6.2.4.c "Prohibited medications" for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study,
* Any ongoing toxicity from prior anti-cancer therapy that is > Grade 1 and/or that is progressing in severity (according to the NCI-CTC AE v4.0), except alopecia,
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2013-03; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure (TTF) | up to 36 months
  TTF is the time to permanent treatment discontinuation due to any cause after randomization in each arm

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 6 months after inclusion
  Proportion of patients with a best overall response of Complete Response (CR) or a Partial Response (PR) at the end of the first 6 cycles, according to RECIST criteria 1.1
Disease Control Rate (DCR) | 6 months after inclusion
  Proportion of patients with a best overall response of Complete Response, Partial Response or Stable Disease at the end of the first 6 cycles, according to RECIST criteria 1.1
Progression-Free Survival (PFS) | up to 36 months
  Time from date of randomization to the date of event defined as the first documented progression under treatment or death due to any cause.
Best response rate | up to 36 months
  Best response observed from date of randomization
Duration of response | up to 36 months
  Time from the first documented response (CR or PR) to the first documented disease progression or death due to any cause, applies only to patients whose best overall response is CR or PR
Overall Survival (OS) | up to 36 months
  Time from date of randomization to the date of death due to any cause
Objective Response Rate (ORR) | 6 months after randomization
  Proportion of patients with a CR or a PR after 6 cycles from randomization.
Disease Control Rate (SDR) | 6 months after randomization
  The proportion of patients with a SD, PR or CR after 6 cycles from randomization.
Safety profile of pazopanib | up to 36 months
  Adverse events (AE) experienced throughout the study and assessed according the NCI-CTC AE version 4.0.
Quality of Life (QoL) | At inclusion, randomization and at the end of pazopanib treatment
  The score obtained at the EORTC Quality of Life Questionnaire C30

OTHER OUTCOMES:
Identification of prognostic biomarkers of clinical outcome. | At inclusion, day 56 and day 168 of treatment (before randomisation)
  To study the correlation between clinical response and biomarkers (serum and tissue).
Tissue expression of Raf-1 kinase inhibitory protein, PAX8, BRAF, Pi3KCA and Ras. | At inclusion, day 56 and day 168 of treatment (before randomization)
  To perform gene expression profiling and to identify potential candidate genes.

CONTACTS AND LOCATIONS:
Overall Officials: Christelle De La Fouchardière, MD, Principal Investigator — Centre Léon Bérard, Lyon
Locations (13):
- France (13):
  - CHU Angers, Angers
  - CHU Bordeaux, Bordeaux
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - CHRU Lille Hôpital Claude Huriez, Lille
  - Centre Leon Berard, Lyon
  - Hôpital de la Timone APHM, Marseille
  - Centre Antoine Lacassagne, Nice
  - Hôpital Saint-Louis APHP, Paris
  - Hôpital de la Pitié Salpêtrière APHP, Paris
  - Institut Jean Godinot, Reims
  - Institut Claudius Régaud, Toulouse
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Bible KC, Suman VJ, Molina JR, Smallridge RC, Maples WJ, Menefee ME, Rubin J, Sideras K, Morris JC 3rd, McIver B, Burton JK, Webster KP, Bieber C, Traynor AM, Flynn PJ, Goh BC, Tang H, Ivy SP, Erlichman C; Endocrine Malignancies Disease Oriented Group; Mayo Clinic Cancer Center; Mayo Phase 2 Consortium. Efficacy of pazopanib in progressive, radioiodine-refractory, metastatic differentiated thyroid cancers: results of a phase 2 consortium study. Lancet Oncol. 2010 Oct;11(10):962-72. doi: 10.1016/S1470-2045(10)70203-5. Epub 2010 Sep 17. PMID 20851682
- [Background] Altorki N, Lane ME, Bauer T, Lee PC, Guarino MJ, Pass H, Felip E, Peylan-Ramu N, Gurpide A, Grannis FW, Mitchell JD, Tachdjian S, Swann RS, Huff A, Roychowdhury DF, Reeves A, Ottesen LH, Yankelevitz DF. Phase II proof-of-concept study of pazopanib monotherapy in treatment-naive patients with stage I/II resectable non-small-cell lung cancer. J Clin Oncol. 2010 Jul 1;28(19):3131-7. doi: 10.1200/JCO.2009.23.9749. Epub 2010 Jun 1. PMID 20516450
- [Background] Billemont B, Medioni J, Taillade L, Helley D, Meric JB, Rixe O, Oudard S. Blood glucose levels in patients with metastatic renal cell carcinoma treated with sunitinib. Br J Cancer. 2008 Nov 4;99(9):1380-2. doi: 10.1038/sj.bjc.6604709. Epub 2008 Oct 7. PMID 18841151
- [Background] Borson-Chazot F, Bardet S, Bournaud C, Conte-Devolx B, Corone C, D'Herbomez M, Henry JF, Leenhardt L, Peix JL, Schlumberger M, Wemeau JL; Expert Group for French Recommendations for the Management of Differentiated Thyroid Carcinomas of Vesicular Origin; Baudin E, Berger N, Bernard MH, Calzada-Nocaudie M, Caron P, Catargi B, Chabrier G, Charrie A, Franc B, Hartl D, Helal B, Kerlan V, Kraimps JL, Leboulleux S, Le Clech G, Menegaux F, Orgiazzi J, Perie S, Raingeard I, Rodien P, Rohmer V, Sadoul JL, Schwartz C, Tenenbaum F, Toubert ME, Tramalloni J, Travagli JP, Vaudrey C. Guidelines for the management of differentiated thyroid carcinomas of vesicular origin. Ann Endocrinol (Paris). 2008 Dec;69(6):472-86. doi: 10.1016/j.ando.2008.10.002. No abstract available. PMID 19137632
- [Background] Brose M. S., et al. Effect of BRAFV600E on response to sorafenib in advanced thyroid cancer patients. J Clin Oncol (meeting Abstracts) 27.15S (2009) : 6002.
- [Background] Carr LL, Mankoff DA, Goulart BH, Eaton KD, Capell PT, Kell EM, Bauman JE, Martins RG. Phase II study of daily sunitinib in FDG-PET-positive, iodine-refractory differentiated thyroid cancer and metastatic medullary carcinoma of the thyroid with functional imaging correlation. Clin Cancer Res. 2010 Nov 1;16(21):5260-8. doi: 10.1158/1078-0432.CCR-10-0994. Epub 2010 Sep 16. PMID 20847059
- [Background] de la Fouchardiere C, Droz JP. Targeted therapies and thyroid cancer: an update. Anticancer Drugs. 2011 Aug;22(7):688-99. doi: 10.1097/CAD.0b013e32834319c7. PMID 21200314
- [Background] Fagin JA, Tuttle RM, Pfister DG. Harvesting the low-hanging fruit: kinase inhibitors for therapy of advanced medullary and nonmedullary thyroid cancer. J Clin Endocrinol Metab. 2010 Jun;95(6):2621-4. doi: 10.1210/jc.2010-0800. No abstract available. PMID 20525911
- [Background] GSK Laboratories. Investigator's Brochure of pazopanib, version 09 dated 25 Jan. 2012.Ref Type: Unpublished Work
- [Background] Gupta-Abramson V, Troxel AB, Nellore A, Puttaswamy K, Redlinger M, Ransone K, Mandel SJ, Flaherty KT, Loevner LA, O'Dwyer PJ, Brose MS. Phase II trial of sorafenib in advanced thyroid cancer. J Clin Oncol. 2008 Oct 10;26(29):4714-9. doi: 10.1200/JCO.2008.16.3279. Epub 2008 Jun 9. PMID 18541894
- [Background] Hutson TE, Davis ID, Machiels JP, De Souza PL, Rottey S, Hong BF, Epstein RJ, Baker KL, McCann L, Crofts T, Pandite L, Figlin RA. Efficacy and safety of pazopanib in patients with metastatic renal cell carcinoma. J Clin Oncol. 2010 Jan 20;28(3):475-80. doi: 10.1200/JCO.2008.21.6994. Epub 2009 Dec 14. PMID 20008644
- [Background] Freedman LS. Tables of the number of patients required in clinical trials using the logrank test. Stat Med. 1982 Apr-Jun;1(2):121-9. doi: 10.1002/sim.4780010204. PMID 7187087
- [Background] Jebreel A, England J, Bedford K, Murphy J, Karsai L, Atkin S. Vascular endothelial growth factor (VEGF), VEGF receptors expression and microvascular density in benign and malignant thyroid diseases. Int J Exp Pathol. 2007 Aug;88(4):271-7. doi: 10.1111/j.1365-2613.2007.00533.x. PMID 17696908
- [Background] Iwamoto FM, Lamborn KR, Robins HI, Mehta MP, Chang SM, Butowski NA, Deangelis LM, Abrey LE, Zhang WT, Prados MD, Fine HA. Phase II trial of pazopanib (GW786034), an oral multi-targeted angiogenesis inhibitor, for adults with recurrent glioblastoma (North American Brain Tumor Consortium Study 06-02). Neuro Oncol. 2010 Aug;12(8):855-61. doi: 10.1093/neuonc/noq025. Epub 2010 Mar 3. PMID 20200024
- [Background] Kaplan, E. L and P. Meier. Nonparametric estimation from incomplete observations. J Am Stat Assoc 53 (1958): 457-81.
- [Background] Kumar R, Knick VB, Rudolph SK, Johnson JH, Crosby RM, Crouthamel MC, Hopper TM, Miller CG, Harrington LE, Onori JA, Mullin RJ, Gilmer TM, Truesdale AT, Epperly AH, Boloor A, Stafford JA, Luttrell DK, Cheung M. Pharmacokinetic-pharmacodynamic correlation from mouse to human with pazopanib, a multikinase angiogenesis inhibitor with potent antitumor and antiangiogenic activity. Mol Cancer Ther. 2007 Jul;6(7):2012-21. doi: 10.1158/1535-7163.MCT-07-0193. PMID 17620431
- [Background] Lan, K. K. G. and D. L. De Mets. Discrete sequential boundaries for clinical trials. Biometrika 70 (1983): 659-63
- [Background] Leboulleux, S., Bastholt, L., and Krause TM. Vandetanib in locally advanced or metastatic differentiated thyroid cancer (papillary or follicular; DTC): a randomized, double-blind phase II trial. International Thyroid Conference;Paris, France; [ Sept 11.16, 2009. Abstr 0C.023.]. 2010. Ref Type: Abstract
- [Background] Monk BJ, Mas Lopez L, Zarba JJ, Oaknin A, Tarpin C, Termrungruanglert W, Alber JA, Ding J, Stutts MW, Pandite LN. Phase II, open-label study of pazopanib or lapatinib monotherapy compared with pazopanib plus lapatinib combination therapy in patients with advanced and recurrent cervical cancer. J Clin Oncol. 2010 Aug 1;28(22):3562-9. doi: 10.1200/JCO.2009.26.9571. Epub 2010 Jul 6. PMID 20606083
- [Background] Nikiforov YE. Thyroid carcinoma: molecular pathways and therapeutic targets. Mod Pathol. 2008 May;21 Suppl 2(Suppl 2):S37-43. doi: 10.1038/modpathol.2008.10. PMID 18437172
- [Background] Pacini F, Castagna MG, Brilli L, Pentheroudakis G; ESMO Guidelines Working Group. Differentiated thyroid cancer: ESMO clinical recommendations for diagnosis, treatment and follow-up. Ann Oncol. 2009 May;20 Suppl 4:143-6. doi: 10.1093/annonc/mdp156. No abstract available. PMID 19454437
- [Background] Prince HM, Honemann D, Spencer A, Rizzieri DA, Stadtmauer EA, Roberts AW, Bahlis N, Tricot G, Bell B, Demarini DJ, Benjamin Suttle A, Baker KL, Pandite LN. Vascular endothelial growth factor inhibition is not an effective therapeutic strategy for relapsed or refractory multiple myeloma: a phase 2 study of pazopanib (GW786034). Blood. 2009 May 7;113(19):4819-20. doi: 10.1182/blood-2009-02-207209. No abstract available. PMID 19423744
- [Background] Ravaud, A., et al. Sunitinib in patients with refractory advanced thyroid cancer: the THYSU phase II trial. J Clin Oncol (Meeting Abstracts) 26.15_suppl (2008): 6058.
- [Background] Ricarte-Filho JC, Ryder M, Chitale DA, Rivera M, Heguy A, Ladanyi M, Janakiraman M, Solit D, Knauf JA, Tuttle RM, Ghossein RA, Fagin JA. Mutational profile of advanced primary and metastatic radioactive iodine-refractory thyroid cancers reveals distinct pathogenetic roles for BRAF, PIK3CA, and AKT1. Cancer Res. 2009 Jun 1;69(11):4885-93. doi: 10.1158/0008-5472.CAN-09-0727. PMID 19487299
- [Background] Schlumberger M. [Papillary and follicular thyroid carcinoma]. Ann Endocrinol (Paris). 2007 Jun;68(2-3):120-8. doi: 10.1016/j.ando.2007.04.004. Epub 2007 Jun 19. French. PMID 17582381
- [Background] Sherman SI, Wirth LJ, Droz JP, Hofmann M, Bastholt L, Martins RG, Licitra L, Eschenberg MJ, Sun YN, Juan T, Stepan DE, Schlumberger MJ; Motesanib Thyroid Cancer Study Group. Motesanib diphosphate in progressive differentiated thyroid cancer. N Engl J Med. 2008 Jul 3;359(1):31-42. doi: 10.1056/NEJMoa075853. PMID 18596272
- [Background] Slamon D,. et al. Pazopanib + Lapatinib is more active than Lapatinib alone : Updated results from a randomized study in patients with first-line ErbB2-positive advanced or metastatic breast cancer [ESMO abstract 139P]. Ann Oncol. 2008c ;19 (supp 8) : viii 64-65.
- [Background] Sleijfer, S., et al. Phase II study of pazopanib (GW786034) in patients (pts) with relapsed or refractory soft tissue sarcoma (STS): EORTC 62043. ASCO Meeting Abstracts 25.18_suppl (2007): 10031.
- [Background] Sternberg CN, Davis ID, Mardiak J, Szczylik C, Lee E, Wagstaff J, Barrios CH, Salman P, Gladkov OA, Kavina A, Zarba JJ, Chen M, McCann L, Pandite L, Roychowdhury DF, Hawkins RE. Pazopanib in locally advanced or metastatic renal cell carcinoma: results of a randomized phase III trial. J Clin Oncol. 2010 Feb 20;28(6):1061-8. doi: 10.1200/JCO.2009.23.9764. Epub 2010 Jan 25. PMID 20100962
- [Background] Soh EY, Duh QY, Sobhi SA, Young DM, Epstein HD, Wong MG, Garcia YK, Min YD, Grossman RF, Siperstein AE, Clark OH. Vascular endothelial growth factor expression is higher in differentiated thyroid cancer than in normal or benign thyroid. J Clin Endocrinol Metab. 1997 Nov;82(11):3741-7. doi: 10.1210/jcem.82.11.4340. PMID 9360534
- [Background] Volante M, Rapa I, Gandhi M, Bussolati G, Giachino D, Papotti M, Nikiforov YE. RAS mutations are the predominant molecular alteration in poorly differentiated thyroid carcinomas and bear prognostic impact. J Clin Endocrinol Metab. 2009 Dec;94(12):4735-41. doi: 10.1210/jc.2009-1233. Epub 2009 Oct 16. PMID 19837916
- [Derived] de la Fouchardiere C, Godbert Y, Dalban C, Illouz F, Wassermann J, Do Cao C, Bardet S, Zerdoud S, Chougnet CN, Zalzali M, Benisvy D, Niccoli P, Digue L, Lamartina L, Schwartz P, Borson Chazot F, Gautier J, Perol D, Leboulleux S; PAZOTHYR investigators. Intermittent versus continuous administration of pazopanib in progressive radioiodine refractory thyroid carcinoma: Final results of the randomised, multicenter, open-label phase II trial PAZOTHYR. Eur J Cancer. 2021 Nov;157:153-164. doi: 10.1016/j.ejca.2021.07.029. Epub 2021 Sep 9. PMID 34509954